CLINICAL TRIAL: NCT00242593
Title: The Effects of Rosiglitazone on Cognition in Patients With MCI
Brief Title: Rosiglitazone Effects on Cognition for Adults in Later Life
Acronym: RECALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH); GlaxoSmithKline (Industry)
Responsible Party: Suzanne Craft, PhD, University of Washington School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0087; 1R01AG025502-01A1 (NIH)
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Mild Cognitive Impairment
Keywords: cognition disorders; Alzheimer's disease; memory
MeSH Terms: conditions — Cognitive Dysfunction; Cognition Disorders; Alzheimer Disease | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): oral rosiglitazone 4 mg twice daily for 18 months
  Interventions: Drug: Rosiglitazone
- B (Placebo Comparator): placebo pill twice daily for 18 months
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — 4 mg twice daily oral rosiglitazone or placebo pill for 18 months
  Other Names: Avandia

SUMMARY:
The purpose of this study is to determine the effects of the insulin-sensitizing medication rosiglitazone on attention and memory skills in older adults with mild cognitive impairment (MCI). The study also will examine the effects of this medication on brain structures that support memory and other thinking abilities, and on biological markers associated with inflammation, insulin resistance, and cardiovascular disease.

DETAILED DESCRIPTION:
The study will examine the effects of the insulin-sensitizing agent rosiglitazone on learning and memory for 120 patients diagnosed with MCI. Participants will be randomized to an 18-month trial of rosiglitazone or placebo, followed by a 2-month washout period. At screening and at treatment month 18, all participants will undergo an oral glucose tolerance test (OGTT) to estimate pre- and post- treatment insulin sensitivity and β-cell function. Cognitive measures and blood samples for biochemical assays will be obtained at baseline, treatment months 6, 12, and 18, and washout (two months after completing treatment).

During treatment, participants will have safety labs drawn and receive physical assessment of any adverse events, changes in health status, or changes in medication; initially these visits will be done at weeks 2 and 4, and then every three months. For months in which a safety visit is not scheduled, telephone monitoring to assess any health concerns will be conducted.

All participants enrolled in the primary study will be approached to participate in an MRI substudy; patients will undergo serial brain MRI before treatment and following 18 months of rosiglitazone or placebo, using three-dimensional T1-weighted images. Comparison of MCI patients receiving rosiglitazone and placebo will be conducted to determine whether the rate of medial temporal lobe (MTL) and whole brain atrophy is altered following treatment.

ELIGIBILITY:
Inclusion Criteria:

* MCI diagnosis: Participants will be diagnosed with MCI by consensus of a team of physicians and neuropsychologists experienced in the diagnosis of MCI, using the Petersen (Petersen, 1999, 2001) criteria for amnestic MCI or multiple domain MCI with amnestic features: a) the presence of subjective memory complaints, evaluated via detailed patient history and informant interview, b) objective verification of memory impairment as measured by neuropsychological tests, c) normal general cognitive function, d) intact or only mildly impaired activities of daily living, and e) absence of dementia per NINCDS/ADRDA and/or DSM-IV criteria

Exclusion Criteria:

The following exclusion criteria will be used, based on initial physical examination, medical history, lab work, and oral glucose tolerance test (OGTT) results:

* Diagnosis of diabetes or other relevant glucoregulatory disorders
* Use of any oral anti-diabetic compounds
* Clinically significant elevations in liver function
* Significant neurological disease that might affect cognition, other than MCI, including Alzheimer's disease, large-vessel stroke, Parkinson's disease, multiple sclerosis, recent severe head injury (loss of consciousness for more than 30 minutes in the past year), or remote head injury resulting in permanent cognitive or neurological sequelae
* History or current evidence of congestive heart failure (CHF)
* History of documented ischemic cardiac disease, i.e., angina, MI, angioplasty, stent, or CABG
* History of cardiac or vascular surgery, or significant arrhythmia within the last year; or planned major intervention such as cardiac surgery or stenting. A history of cardiac surgery for non-ischemic indications (i.e., valve repair or replacement) greater than one year prior to enrollment is not exclusionary if all other criteria are met
* Significant ECG abnormalities including heart rate less than 50 or greater than 100 beats per minute (dependent upon the individual's general health); any previously unrecognized arrhythmia requiring further intervention
* Significant peripheral edema at the time of screening
* Significant medical illness or organ failure, including but not limited to renal disease, hepatic disease, and unstable cardiac disease
* Regular current use of antipsychotic, anticonvulsive, anxiolytic, or sedative medications; antidepressant medications are not exclusionary, provided the individual does not have current major depression
* A current diagnosis of major depression or other significant psychiatric comorbidity
* Clinically significant anemia at the time of screening
* Fasting triglyceride level greater than 400
* Fasting glucose 125 or greater, or two-hour glucose value greater than 199 during the OGTT; participants will be notified if their fasting blood sugar (monitored every 3 months) exceeds 125, and they will be withdrawn from further participation if their fasting blood sugar exceeds 125 for two consecutive months
* For the MRI substudy, additional exclusion criteria include 1) previous exposure to work involving the cutting or grinding of metal, 2) the presence of a pacemaker, aneurysm clip, or other implanted metal device that would prohibit MRI procedures, and 3) significant history of claustrophobia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive measures: delayed list recall, Stroop Interference test | every 6 months for 18 months, again 2 at months post-treatment (20 months)
Biological outcomes: plasma insulin, IDE, AB40, AB42, inflammatory cytokines, and F2-isoprostanes | every 6 months for 18 months, again 2 at months post-treatment (20 months)
MRI outcome: Whole brain and medial temporal lobe atrophy rate | baseline and 18 months

SECONDARY OUTCOMES:
Cognitive measures: ADAS-cog total score, story recall verbal fluency, paired associate learning, SOPT, rating scales | every 6 months for 18 months, again 2 at months post-treatment (20 months)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Craft, PhD, Principal Investigator — University of Washington/VA Puget Sound Health Care System
Locations (3):
- United States (3):
  - Banner Alzheimer Institute, Phoenix, Arizona
  - UCLA Alzheimer's Disease Center, Los Angeles, California
  - University of Washington/VA Puget Sound Health Care System, Seattle/Tacoma, Washington

REFERENCES:
- [Background] Goldstein BJ. Rosiglitazone. Int J Clin Pract. 2000 Jun;54(5):333-7. PMID 10954962
- [Background] Mudaliar S, Henry RR. New oral therapies for type 2 diabetes mellitus: The glitazones or insulin sensitizers. Annu Rev Med. 2001;52:239-57. doi: 10.1146/annurev.med.52.1.239. PMID 11160777
- [Background] Lopez OL, Jagust WJ, Dulberg C, Becker JT, DeKosky ST, Fitzpatrick A, Breitner J, Lyketsos C, Jones B, Kawas C, Carlson M, Kuller LH. Risk factors for mild cognitive impairment in the Cardiovascular Health Study Cognition Study: part 2. Arch Neurol. 2003 Oct;60(10):1394-9. doi: 10.1001/archneur.60.10.1394. PMID 14568809
- [Background] Gasparini L, Gouras GK, Wang R, Gross RS, Beal MF, Greengard P, Xu H. Stimulation of beta-amyloid precursor protein trafficking by insulin reduces intraneuronal beta-amyloid and requires mitogen-activated protein kinase signaling. J Neurosci. 2001 Apr 15;21(8):2561-70. doi: 10.1523/JNEUROSCI.21-08-02561.2001. PMID 11306609
- [Background] Watson GS, Craft S. The role of insulin resistance in the pathogenesis of Alzheimer's disease: implications for treatment. CNS Drugs. 2003;17(1):27-45. doi: 10.2165/00023210-200317010-00003. PMID 12467491